CLINICAL TRIAL: NCT02322411
Title: Effects of Device-Facilitated Isometric Progressive Resistance Oropharyngeal (I-PRO) Therapy on Dysphagia Related Outcomes in Patients Post-stroke
Brief Title: Effects of Oropharyngeal Strengthening on Dysphagia in Patients Post-stroke
Acronym: StrokeStrong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0747; A534255 (Other: UW, Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW, Madison)
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Stroke; Deglutition; Deglutition disorders; Resistance training
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Compensatory (Active Comparator): This group will receive standard swallowing intervention, which is identified by the SLP as appropriate to treat the patient's dysphagia and is common clinical practice. Their therapy may include: 1) modifying their foods and fluids; 2) changing their posture when they eat or drink; or 3) having them eat more slowly or in a quiet environment to make swallowing easier and safer. These compensatory approaches will ensure safety while swallowing foods and fluids. Range of motion, vocal exercises, and other oromotor exercises, such as the Shaker Exercise, as well as any other potential strengthening regimens for swallowing or speech will be delayed until subjects have completed participation.
  Interventions: Behavioral: Compensatory approaches
- I-PRO + compensatory (Experimental): The Device-Facilitated Isometric Progressive Resistance Oropharyngeal (D-F I-PRO) intervention will be completed using the SwallowSTRONG® device. Tongue press exercises consist of pressing the tongue against the sensors located along the hard palate. Isometric exercises will focus on the anterior and posterior sensor. Subjects will take the SwallowStrong® device home with them and will complete 20 repetitions of the exercise (10 repetitions at the front sensor; 10 repetitions at the back sensor), three times per day on three days per week for twelve weeks.
  Interventions: Device: Isometric Progressive Resistance Oropharyngeal Therapy; Behavioral: Compensatory approaches

INTERVENTIONS:
Device: Isometric Progressive Resistance Oropharyngeal Therapy — Isometric Progressive Resistance Oropharyngeal Therapy is an approach to oropharyngeal strengthening. This particular use of I-PRO therapy will be facilitated by the Swallow Strong device.
  Other Names: SwallowStrong device
  Arms: I-PRO + compensatory
Behavioral: Compensatory approaches

SUMMARY:
The overall goal of this randomized controlled pilot study is to characterize effects of SwallowSTRONG® Device-Facilitated Isometric Progressive Resistance Oropharyngeal (DF I-PRO) therapy in a dose response framework on swallowing-related outcomes in a group of unilateral ischemic stroke patients. These results will be used to determine adequate sample size in order to support a larger clinical trial focused on the efficacy of this therapy approach for improving swallowing safety. The first aim is to determine differences in swallowing physiology and bolus flow measures a) between a group of unilateral ischemic stroke subjects undergoing SwallowSTRONG® DF I-PRO therapy and controls and b) between 8 and 12 weeks of treatment. The second aim is to examine changes in level of oral intake and swallowing quality of life in post-stroke patients undergoing DF I-PRO therapy as compared to a control group and as they relate to treatment duration response at 8 weeks and 12 weeks. The third aim is to evaluate effects of DF I-PRO therapy on overall health status reflected by the number of pneumonia diagnoses and overall hospital readmission rates in post-stroke subjects undergoing DF I-PRO therapy compared to controls.

DETAILED DESCRIPTION:
Dysphagia is estimated to occur in up to 76% of acute stroke patients1,2 and by 2030 the prevalence of stroke is estimated to rise by 21%.3 Serious health complications may result from the presence of dysphagia following stroke, including the development of aspiration pneumonia, malnutrition, and mortality.4-6 Developing pneumonia post-stroke results in a significantly increased relative risk (2.99) of death within 30 days of hospital discharge.1 Compensatory approaches to intervention, including postures or diet modification, are commonly used but do not enact lasting change in swallowing function. Early and intensive therapy approaches are suggested for attainment of optimal swallowing outcomes.7 The tongue is the primary propulsive force for movement of the bolus through the oral cavity and pharynx and into the cervical esophagus during swallowing. Patients post-stroke demonstrate lower than normal maximum isometric lingual pressures, measured as pressures produced when the tongue is pushed as hard as possible against the palate.2 Progressive resistance training for the tongue and related oropharyngeal musculature has been shown to improve swallow physiology and quality of life for patients post-stroke.8 Previous studies have examined Isometric Progressive Resistance Oropharyngeal (I-PRO) therapy facilitated by the Iowa Oral Pressure Instrument (IOPI) for lingual strengthening. The recently developed SwallowSTRONG® device consists of a customized, adjustable mouthpiece that provides pressure readings from embedded sensors allowing for consistent tongue placement, immediate knowledge of performance levels, and automatic calculation of therapeutic strengthening targets. Results from a federally-funded Department of Veterans Affairs Clinical Demonstration Program that employed use of device-facilitated (DF) I-PRO therapy showed improved swallowing-related outcomes in a group of patients with oropharyngeal dysphagia resulting from a variety of medical etiologies.9 The effects of this therapy approach on various aspects of swallowing function and health status in a group of post-stroke patients have yet to be examined. In addition, ideal treatment duration for use with stroke patients is unknown.

The long term goal of this work is to develop more effective, evidence-based treatments that improve overall health status related to swallowing-specific changes for patients with dysphagia. The preliminary group data generated will provide the basis for a line of work dedicated to determination of effective treatments for patients post-stroke.

Specific Aims include: 1) determine differences in swallowing physiology and bolus flow measures a) between a group of unilateral ischemic stroke subjects undergoing DF I-PRO therapy and a control group and b) between two durations of treatment (8 and 12 weeks); 2) examine changes in level of oral intake and swallowing quality of life in post-stroke patients undergoing I-PRO therapy as compared to a control group and as they relate to treatment duration response at 8 weeks and 12 weeks; and 3) evaluate effects of DF I-PRO therapy on overall health status reflected by the number of pneumonia diagnoses and overall hospital readmission rates in post-stroke subjects undergoing DF I-PRO therapy compared to controls.

In order to address these aims, thirty patients who have suffered unilateral ischemic stroke will be recruited. Subjects will be randomized to receive either 1) 12 weeks of DF I-PRO therapy plus compensatory treatment or 2) compensatory treatment only. Assessments will take place at baseline, 8 and 12 weeks. The primary outcome measure will be changes in maximum isometric tongue pressures. Details regarding specific outcomes most influenced by this approach and dose response effects will inform the clinical practice of Speech-Language Pathologists and facilitate strengthening regimens to become more standard for the treatment of stroke related dysphagia.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of unilateral ischemic strokes by attending physician (according to the National Institute of Health Stroke Scale (NIHSS))
2. within 6 months of acute stroke diagnosis
3. a score of 3 or higher on the Penetration-Aspiration scale OR a score of 2 on the Residue scale at any location (oral cavity, valleculae, or pharynx) that is instrumentally documented by a participating SLP during a standardized videofluoroscopic swallowing study
4. between the ages of 21 and 95
5. ability to perform the strengthening protocol independently or with the assistance of a caregiver
6. physician approval of medical stability to participate
7. decision-making capacity to provide informed consent (confirmed through discussion with the subject's primary physician)
8. phone access
9. ability to return to the clinic for required follow-up appointments.

Exclusion Criteria:

1. degenerative neuromuscular disease
2. prior or current diagnosis of bilateral or hemorrhagic stroke
3. prior surgery to the head and neck region that would affect muscles involved in swallowing
4. history of radiotherapy or chemotherapy to the head and neck
5. patient unable to complete the exercise program
6. taking medications that depress the central nervous system
7. allergy to barium (used in videofluoroscopic swallowing assessment)
8. currently pregnant.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Pulia, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Krekeler BN, Yee J, Kurosu A, Osman F, Pena-Chavez R, Leverson G, Young B, Sattin J, Knigge M, Thibeault S, Rogus-Pulia N. Effects of Device-Facilitated Lingual Strengthening Therapy on Dysphagia Related Outcomes in Patients Post-Stroke: A Randomized Controlled Trial. Dysphagia. 2023 Dec;38(6):1551-1567. doi: 10.1007/s00455-023-10583-0. Epub 2023 May 17. PMID 37195518

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants were consented to the study, 14 randomized to the compensatory arm, 16 to the I-PRO + compensatory arm. 1 participant in the compensatory arm withdrew after baseline residue analysis only (this participant's data is reported at baseline in the Residue Analysis Outcome Measure)
Groups:
- Compensatory: This group will receive standard swallowing intervention, which is identified by the SLP as appropriate to treat the patient's dysphagia and is common clinical practice. Their therapy may include: 1) modifying their foods and fluids; 2) changing their posture when they eat or drink; or 3) having them eat more slowly or in a quiet environment to make swallowing easier and safer. These compensatory approaches will ensure safety while swallowing foods and fluids. Range of motion, vocal exercises, and other oromotor exercises, such as the Shaker Exercise, as well as any other potential strengthening regimens for swallowing or speech will be delayed until subjects have completed participation.
  Compensatory approaches
- I-PRO + Compensatory: The Device-Facilitated Isometric Progressive Resistance Oropharyngeal (D-F I-PRO) intervention will be completed using the SwallowSTRONG® device. Tongue press exercises consist of pressing the tongue against the sensors located along the hard palate. Isometric exercises will focus on the anterior and posterior sensor. Subjects will take the SwallowStrong® device home with them and will complete 20 repetitions of the exercise (10 repetitions at the front sensor; 10 repetitions at the back sensor), three times per day on three days per week for twelve weeks.
  Isometric Progressive Resistance Oropharyngeal Therapy: Isometric Progressive Resistance Oropharyngeal Therapy is an approach to oropharyngeal strengthening. This particular use of I-PRO therapy will be facilitated by the Swallow Strong device.
  Compensatory approaches
Period: Overall Study
Arm/Group | Compensatory | I-PRO + Compensatory
Started | 14 | 16
Randomized | 14 | 16
All Baseline Measures Analyzed | 13 | 16
Completed | 9 | 9
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 4 | 7
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Compensatory | I-PRO + Compensatory | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (15.5) | 68.9 (12.0) | 70.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 16 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Lingual Pressures (Changes in the One Repetition Maximum Isometric Lingual Pressures)
Description: Changes in the one repetition maximum isometric lingual pressures measured at the front and back sensors of the device
Time Frame: After 8 weeks and 12 weeks
Population: Front/Back Lingual Pressure at 8 weeks and 12 weeks - 6 subjects for Compensatory group Front/Back Lingual Pressure at 8 weeks - 8 subjects for I-PRO group Front/Back Lingual Pressure at 12 weeks - 6 subjects for I-PRO group
Measure: Mean (Standard Deviation); unit: hPa
Arm/Group | Compensatory | I-PRO + Compensatory
Number analyzed (Participants) | 13 | 16
hPa
  Front Lingual Pressure at 8 weeks: number analyzed (Participants) | 6 | 8
  Front Lingual Pressure at 8 weeks | 83.3 (71.9) | 239.6 (123.0)
  Front Lingual Pressure at 12 weeks: number analyzed (Participants) | 6 | 6
  Front Lingual Pressure at 12 weeks | 129.8 (108.0) | 386.3 (229.9)
  Back Lingual Pressure at 8 weeks: number analyzed (Participants) | 6 | 8
  Back Lingual Pressure at 8 weeks | 31.5 (52.6) | 127.6 (158.9)
  Back Lingual Pressure at 12 weeks: number analyzed (Participants) | 6 | 6
  Back Lingual Pressure at 12 weeks | 50.05 (55.6) | 131.4 (118.9)

2. Secondary Outcome: Percent Residue
Description: Measurement of Residue
Time Frame: baseline, 8 and 12 weeks
Population: Not all participants had analyzable swallow studies, one participant in the Compensatory Arm withdrew from the study after the baseline residue analysis.
Measure: Mean (Standard Deviation); unit: Percent Residue
Arm/Group | Compensatory | I-PRO + Compensatory
Number analyzed (Participants) | 14 | 14
Percent Residue
  Baseline Total Residue | 9.12 (8.39) | 10.20 (8.54)
  8-Week Total Residue: number analyzed (Participants) | 7 | 6
  8-Week Total Residue | 7.14 (5.22) | 7.12 (4.67)
  12-Week Total Residue: number analyzed (Participants) | 4 | 4
  12-Week Total Residue | 5.65 (3.27) | 7.55 (4.27)

3. Secondary Outcome: Swallowing-related Pressures (Videofluoroscopic Swallow Study)
Description: Pressures will be measured while the subject is swallowing during the videofluoroscopic swallow study
Time Frame: After 8 and 12 weeks
Population: Data for this secondary outcome measure was not collected as the equipment stopped working at the start of the study. The study team did not have the resources to purchase new equipment to collect these data.
Arm/Group | Compensatory | I-PRO + Compensatory
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Dysphagia-related Quality of Life Scores (SWAL-QOL)
Description: A quality of life questionnaire related to swallowing. The scores range from 0-100, and a higher score indicates a higher quality of life related to swallowing.
Time Frame: After 8 weeks and 12 weeks
Population: SWAL-QOL score at 8 weeks - 9 subjects for I-PRO group SWAL-QOL score at 12 weeks - 6 subjects for I-PRO group SWAL-QOL score at 8 weeks - 7 subjects for compensatory group SWAL-QOL score at 12 weeks - 7 subjects for compensatory group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory | I-PRO + Compensatory
Number analyzed (Participants) | 13 | 16
score on a scale
  SWAL-QOL score at 8 weeks: number analyzed (Participants) | 7 | 9
  SWAL-QOL score at 8 weeks | 86.0 (14.6) | 85.5 (8.5)
  SWAL-QOL score at 12 weeks: number analyzed (Participants) | 7 | 6
  SWAL-QOL score at 12 weeks | 88.9 (5.0) | 86.3 (8.1)

5. Secondary Outcome: Functional Oral Intake Scale (FOIS) Scores
Description: FOIS scores reflect level of nutritional intake. Scores range from 1 to 7, with 1 being nothing by mouth and with 7 indicating a diet with no restrictions. Qualitative assessment via interview. Range of final scores is between 1 and 7. Average scores of each arm reported at 8 and 12 weeks.
Time Frame: After 8 weeks and 12 weeks
Population: FOIS score at 8 weeks - 9 subjects for I-PRO group FOIS score at 8 weeks - 10 subjects for compensatory group FOIS score at 12 weeks - 8 subjects for I-PRO group FOIS score at 12 weeks - 6 subjects for compensatory group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compensatory | I-PRO + Compensatory
Number analyzed (Participants) | 13 | 16
score on a scale
  FOIS score at 8 weeks: number analyzed (Participants) | 10 | 9
  FOIS score at 8 weeks | 5.6 (1.9) | 6.8 (0.4)
  FOIS score at 12 weeks: number analyzed (Participants) | 6 | 8
  FOIS score at 12 weeks | 5.8 (1.2) | 6.9 (0.4)

6. Secondary Outcome: Pneumonia Diagnoses (Number of Pneumonia Diagnoses)
Description: The number of pneumonia diagnoses within 9 months following completion of the program will be compared to the same pre-enrollment period.
Time Frame: up to 9 months
Measure: Number; unit: incidences of pneumonia
Arm/Group | Compensatory | I-PRO + Compensatory
Number analyzed (Participants) | 13 | 16
incidences of pneumonia | 0 | 0

7. Secondary Outcome: Hospital Admissions (Number of Hospital Admissions and Readmissions)
Description: The number of hospital admissions and readmissions within 9 months following completion of the program will be compared to the same pre-enrollment period.
Time Frame: up to 9 months
Measure: Number; unit: hospital admissions
Arm/Group | Compensatory | I-PRO + Compensatory
Number analyzed (Participants) | 13 | 16
hospital admissions
  Admissions pre-enrollment | 1 | 0
  Admission post-enrollment | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Compensatory | I-PRO + Compensatory
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT02322411/Prot_SAP_000.pdf